CLINICAL TRIAL: NCT01567137
Title: Using Magnetic Resonance Techniques to Improve the Characterisation and Localisation of Breast Cancer
Brief Title: MR Characterisation/Localisation of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Principal Investigator, NdeSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: CCR 2995 07/H0806/85
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: To determine the accuracy of multi-functional magnetic resonance (MR) in detecting, localising and characterising satellite lesions in relation to an index breast tumour in order to improve definition of clinical target volume after local excision.

Hypothesis: Pre-operative multi-functional MR has high sensitivity and specificity for localising unsuspected multifocal and multicentric lesions in women diagnosed with early breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven invasive ductal carcinoma of the breast
* Unifocal disease
* Patient proceeding to mastectomy

Exclusion Criteria:

* Multifocal disease
* Previous surgery to ipsilateral breast
* Neoadjuvant chemotherapy
* Ferromagnetic implants
* Claustrophobia
* Cup size DD or greater

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with confirmed breast cancer
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of MR techniques in detecting histopathologically-identified multifocal and multicentric lesions | 4 years
  Sensitivity of the MR technique in detecting histopathologically-identified multifocal/centric pre-invasive/invasive disease will be calculated (with 95% confidence intervals)from positive or negative correlates.

SECONDARY OUTCOMES:
Closeness of agreement between MR techniques and histopathology in localising satellite lesions relative to the index tumour. | 4 years
  Distance & distribution of lesions from reference tumour will be plotted and correlated with distances and signal characteristics seen on multifunctional MR.
  Pre-op MRI volume will be plotted against histopathological dimensions and examined for agreement between the two methods.
  Paired Wilcoxon signed-rank tests will be used to test for systematic differences between MRI and pathology measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom